CLINICAL TRIAL: NCT03617510
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Multiple-dose,Dose-escalated Phase I Clinical Study Trial to Evaluate the Tolerance and Pharmacokinetics of Felbinac Trometamol Injection in Healthy Subjects
Brief Title: A Phase I Clinical Study Trial of Felbinac Trometamol Injection in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BALF-PAIN-1002
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Pain
Keywords: Tolerance; Pharmacokinetic characteristics
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group1 (Experimental): Generic name:Felbinac Trometamol Injection;Placebo:normal saline Dosage form:Injection Dosage:47.13mg Volume:2.00ml Frequency:Multi-dose after single-dose Duration:5 days A total of 12 subjects,10 received the test drug and 2 received the placebo.
  Interventions: Drug: Felbinac Trometamol Injection; Drug: Placebos
- group2 (Experimental): Generic name:Felbinac Trometamol Injection;Placebo:normal saline Dosage form:Injection Dosage:94.25mg Volume:4.00ml Frequency:Multi-dose after single-dose Duration:5 days A total of 12 subjects,10 received the test drug and 2 received the placebo.
  Interventions: Drug: Felbinac Trometamol Injection; Drug: Placebos
- group3 (Experimental): Generic name:Felbinac Trometamol Injection;Placebo:normal saline Dosage form:Injection Dosage:188.50mg Volume:8.00ml Frequency:Multi-dose after single-dose Duration:5 days A total of 12 subjects,10 received the test drug and 2 received the placebo.
  Interventions: Drug: Felbinac Trometamol Injection; Drug: Placebos
- group4 (Experimental): Generic name:Felbinac Trometamol Injection;Placebo:normal saline Dosage form:Injection Dosage:259.16mg Volume:11.00ml Frequency:Multi-dose after single-dose Duration:5 days A total of 12 subjects,10 received the test drug and 2 received the placebo.
  Interventions: Drug: Felbinac Trometamol Injection; Drug: Placebos

INTERVENTIONS:
Drug: Felbinac Trometamol Injection — Felbinac Trometamol Injection will be infused IV in 100 mL normal saline,in a 30-minute period using a programmable pump.Three days after the single dose,the drug was given 7 times,3 times/day,once every 8 hours. It means the drug was given 3 times on D3 and D4,once on D5.
  Other Names: 4-Biphenylacetic Acid
Drug: Placebos — Normal saline will be infused IV in 100 mL normal saline,in a 30-minute period using a programmable pump.Three days after the single dose,the Placebo was given 7 times,3 times/day,once every 8 hours.It means the Placebo was given 3 times on D3 and D4,once on D5.
  Other Names: normal saline

SUMMARY:
1. To evaluate the tolerances of healthy subjects treated with Felbinac Trometamol Injection on multiple dose and single dose
2. To evaluate the pharmacokinetic characteristics in healthy subjects treated with Felbinac Trometamol Injection on multiple dose and single dose
3. To provide the basis for the dose for the follow-up clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions;
2. Be able to complete the research according to the clinical trial protocol;
3. Subjects have no pregnancy plan within the next 6 months and voluntarily take effective contraceptive measures;
4. Male and female subjects between 18 and 45 years (inclusive) of age;
5. Male subjects weighing no less than 50 kg, female subjects weighing no less than 45 kg.Body Mass Index (BMI) 18 to 28 kg/m2 (inclusive);
6. Physical examination, vital signs normal or no clinical significance.

Exclusion Criteria:

1. Someone smoking more than 5 pieces per day within the 3 months before the trial ；
2. Allergies, such as allergies to two or more drugs, food and pollen, or known to the drug component or ethylbenzene ethyl acetate allergy;
3. Having a history of drug and / or alcohol abuse (14 units of alcohol per week: 1 units = beer 285 mL, or 25 mL of spirits, or 100 mL of wine)；
4. Blood donation or extensive blood loss (> 400 mL) within three months of the use of the study drug;
5. Taked any drug that changes liver enzyme activity 28 days prior to the use of the study drug;
6. Taked any prescription, OTC drugs, any vitamin products or herbs within 14 days prior to the use of the study drug;
7. Two weeks before the trial took a special diet (including dragon fruit, mango, grapefruit, and / or rich in xanthine diet, etc.) or strenuous exercise, and other avtivites that affect drug absorption, distribution, metabolism, excretion and so on;
8. Combined with the following CYP3A4, p-gp or Bcrp inhibitors or inducers, such as itraconazole, ketoconazole or dronedarone;
9. There have been significant changes in diet or exercise habits recently;
10. Taked research drugs within three months prior to the use of the study drug or participating in any drug clinical trial;
11. Suffering from any increased risk of hemorrhagic disease, such as hemorrhoids, acute gastritis or stomach and duodenal ulcers;
12. ECG has clinical significance;
13. Female subjects are in lactation or serum pregnancy test are positive during screening or during the test.
14. Clinical laboratory tests are abnormal and have clinical significance, or other clinical findings showing clinically significant diseases (including but not limited to gastrointestinal, renal, liver, nerves, blood, endocrine, neoplasms, lungs, immunizations, mental or heart Cerebrovascular disease);
15. hepatitis (including hepatitis B and hepatitis C), AIDS, syphilis screening test positive;
16. Acute disease occurs before screening or using test drug;
17. Taking chocolate, any caffeine, or xanthine-rich food or drink at least 48 hours prior to the use of the study drug;
18. Taking any alcoholic products within 24 hours prior to the use of the study drug;
19. Alcohol or drug screening positive or drug abuse history over the past five years or 3 months before the trial used by drug users.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Tolerance evaluation index | up to 96.5 hours after mutil-dose
  percent of subjects with adverse reactions

SECONDARY OUTCOMES:
Tmax | up to 96.5 hours after mutil-dose
  The amount of time that a drug is present at the maximum concentration in serum.
Peak Plasma Concentration (Cmax) | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
t1/2 | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
Vd | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
Mean residence time (MRT) parameter. | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
Ke | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
Area under the plasma concentration versus time curve (AUC0-∞) | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
AUC0-48 | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample
Ae0-48 | up to 96.5 hours after mutil-dose
  The PK parameters of the urine and the stool sample
AUC0-last | up to 96.5 hours after mutil-dose
  The PK parameters of the plasma sample

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No